CLINICAL TRIAL: NCT01164033
Title: An Open-Label, Randomized 3-Way Crossover, Study to Examine the Food-Effect on Pharmacokinetics of the Current Formulation and Relative Bioavailability of Two New Formulations for RO5045337 in Patients With Solid Tumors Including Lymphoma
Brief Title: A Study of RO5045337 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NP25299
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (4):
- A (Active Comparator)
  Interventions: Drug: RO5045337
- B (Experimental)
  Interventions: Drug: RO5045337
- C (Experimental)
  Interventions: Drug: RO5045337
- D (Experimental)
  Interventions: Drug: RO5045337

INTERVENTIONS:
Drug: RO5045337 — single oral dose

SUMMARY:
This open-label, randomized, cross-over study will evaluate the effect of food on the pharmacokinetics of single oral doses of RO5045337 in patients with solid tumors. The anticipated time on study treatment is 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Histologically confirmed solid tumor
* Life expectancy of >/=12 weeks
* ECOG performance status of 0 or 1
* Adequate bone marrow, renal and hepatic function

Exclusion Criteria:

* Patients receiving any other investigational agent or therapy administered with the intention to treat their malignancy within 28 days prior to study start
* Patients with pre-existing gastro-intestinal disorder
* Patients with uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Examination of potential food-effect on pharmacokinetics of RO5045337 | 3 weeks
Evaluation of relative bioavailability of RO5045337 | 3 weeks

SECONDARY OUTCOMES:
Evaluation of safety and tolerability of RO5045337 | 3 weeks
Evaluation of pharmacodynamics and biomarkers | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (5):
  - Scottsdale, Arizona
  - Kansas City, Kansas
  - Kensignton, Maryland
  - Dallas, Texas
  - San Antonio, Texas

REFERENCES:
- [Derived] Patnaik A, Tolcher A, Beeram M, Nemunaitis J, Weiss GJ, Bhalla K, Agrawal M, Nichols G, Middleton S, Beryozkina A, Sarapa N, Peck R, Zhi J. Clinical pharmacology characterization of RG7112, an MDM2 antagonist, in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2015 Sep;76(3):587-95. doi: 10.1007/s00280-015-2830-8. Epub 2015 Jul 26. PMID 26210682